CLINICAL TRIAL: NCT02937207
Title: Study on the Treatment of Bronchial Asthma With Traditional Chinese Medicine
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai University of Traditional Chinese Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: LH20161013
Record Dates: First submitted 2016-10-14; First posted 2016-10-18 (Estimated); Last update posted 2020-02-26 (Actual); Status verified 2019-12

CONDITIONS: Bronchial Asthma
Keywords: Bronchial Asthma; Traditional Chinese Medicine
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Hanxiao treatment group (Experimental): 36 patients of exacerbation group belongs to cold type of asthma will take Ke Chuan Liu Wei Mixture oral therapy twice everyday for 14 days and background therapy of ICS and beta2-agonist.
  Interventions: Drug: Ke Chuan Liu Wei Mixture
- Hanxiao control group (Placebo Comparator): 36 patients of exacerbation group belongs to cold type of asthma will take Ke Chuan Liu Wei Mixture placebo oral therapy twice everyday for 14 days and background therapy of ICS and beta2-agonist.
  Interventions: Drug: Ke Chuan Liu Wei Mixture placebo
- Fengtanxiao treatment group (Experimental): 36 patients of exacerbation group belongs to wind phlegm type of asthma will take Chuan Xiong Ping Chuan Mixture and Xie Wu Capsule oral therapy twice everyday for 14 days and background therapy of ICS and beta2-agonist.
  Interventions: Drug: Chuan Xiong Ping Chuan Mixture; Drug: Xie Wu Capsule
- Fengtanxiao control group (Placebo Comparator): 36 patients of exacerbation group belongs to wind phlegm type of asthma will take Chuan Xiong Ping Chuan Mixture placebo and Xie Wu Capsule placebo oral therapy twice everyday for 14 days and background therapy of ICS and beta2-agonist.
  Interventions: Drug: Chuan Xiong Ping Chuan Mixture placebo; Drug: Xie Wu Capsule placebo
- Rexiao treatment group (Experimental): 36 patients of exacerbation group belongs to hot type of asthma will take Dan Ma Jia Tablet oral therapy thrice everyday for 14 days and background therapy of ICS and beta2-agonist.
  Interventions: Drug: Dan Ma Jia Tablet
- Rexiao control group (Placebo Comparator): 36 patients of exacerbation group belongs to hot type of asthma will take Dan Ma Jia Tablet placebo oral therapy thrice everyday for 14 days and background therapy of ICS and beta2-agonist.
  Interventions: Drug: Dan Ma Jia Tablet placebo
- Xuxiao treatment group (Experimental): 36 patients of remission phase of Yang deficiency of asthma will take Zhi Chuan Capsule and Bu Shen Na Qi Granule oral therapy thrice everyday for 14 days and background therapy of ICS and beta2-agonist.
  Interventions: Drug: Zhi Chuan Capsule; Drug: Bu Shen Na Qi Granule
- Xuxiao control group (Placebo Comparator): 36 patients of remission phase of Yang deficiency of asthma will take Zhi Chuan Capsule placebo and Bu Shen Na Qi Granule placebo oral therapy thrice everyday for 14 days and background therapy of ICS and beta2-agonist.
  Interventions: Drug: Zhi Chuan Capsule placebo; Drug: Bu Shen Na Qi Granule placebo

INTERVENTIONS:
Drug: Ke Chuan Liu Wei Mixture — Experience formula of famous traditional Chinese professor Yingen Wu
  Other Names: Ke Chuan Liu Wei He Ji
  Arms: Hanxiao treatment group
Drug: Chuan Xiong Ping Chuan Mixture — Experience formula of famous traditional Chinese professor Changrong Shao
  Other Names: Chuan Xiong Ping Chuan He Ji
  Arms: Fengtanxiao treatment group
Drug: Xie Wu Capsule — Experience formula of famous traditional Chinese professor Jianhua Hu
  Other Names: Xie Wu Jiao Nang
  Arms: Fengtanxiao treatment group
Drug: Dan Ma Jia Tablet — Experience formula of famous traditional Chinese professor Xiaopu Xu
  Other Names: Dan Ma Jia Pian
  Arms: Rexiao treatment group
Drug: Zhi Chuan Capsule — Experience formula of famous traditional Chinese professor Yingen Wu
  Other Names: Zhi Chuan Jiao Nang
  Arms: Xuxiao treatment group
Drug: Bu Shen Na Qi Granule — Experience formula of famous traditional Chinese professor Changrong Shao
  Other Names: Bu Shen Na Qi Ke Li
  Arms: Xuxiao treatment group
Drug: Ke Chuan Liu Wei Mixture placebo — Low dose combination for treating prescription of Ke Chuan Liu Wei Mixture
  Other Names: placebo
  Arms: Hanxiao control group
Drug: Chuan Xiong Ping Chuan Mixture placebo — Low dose combination for treating prescription of Chuan Xiong Ping Chuan Mixture
  Other Names: placebo
  Arms: Fengtanxiao control group
Drug: Xie Wu Capsule placebo — Low dose combination for treating prescription of Xie Wu Capsule
  Other Names: placebo
  Arms: Fengtanxiao control group
Drug: Dan Ma Jia Tablet placebo — Low dose combination for treating prescription of Dan Ma Jia Tablet
  Other Names: placebo
  Arms: Rexiao control group
Drug: Zhi Chuan Capsule placebo — Low dose combination for treating prescription of Zhi Chuan Capsule
  Other Names: placebo
  Arms: Xuxiao control group
Drug: Bu Shen Na Qi Granule placebo — Low dose combination for treating prescription of Bu Shen Na Qi Granule
  Other Names: placebo
  Arms: Xuxiao control group

SUMMARY:
The purpose of this study is to evaluate the clinical efficacy of traditional Chinese medicine in the treatment of asthma, and to promote the application in community hospitals.

DETAILED DESCRIPTION:
Asthma is a serious global health problem and has increasing prevalence in many countries.Although asthma symptoms can be controlled by drug treatment to a large extent, there is still inadequate.Traditional Chinese medicine has a long history of treating asthma, and has a good clinical curative effect.The purpose of this study is to evaluate the clinical efficacy of traditional Chinese medicine in the treatment of asthma, and to promote the application in community hospitals. This could constitute a significant advance in asthma management.

In this study, the investigators recruited patients with asthma exacerbation and remission stage, and gave the corresponding western medicine background treatment and traditional Chinese medicine treatment program.Participants will undergo a physical examination, lung function, blood and sputum collection.

Exacerbation group belongs to cold type of asthma patients will take Ke Chuan Liu Wei Mixture, wind phlegm type of asthma patients will take Chuan Xiong Ping Chuan Mixture and Xie Wu Capsule，and hot type of asthma patients will take Dan Ma Jia Tablet for 14 days treatment, while the 3 control groups were given 3 corresponding placebo treatment for a total of 14 days.

Remission phase of Yang deficiency patients in treatment group will take Zhi Chuan Capsule and Bu Shen Na Qi Granule, and in control group received a placebo treatment for a total of 60 days.

Study visits will occur for 7 days of exacerbation group and 1 year for remission group. Questionnaires to assess asthma control will be completed during study of asthma at exacerbation stage within 44 days and on remission period within 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients had positive bronchodilator reversibility test or positive bronchial challenge test or more than 50 parts per billion of FENO before
* Number of months without control between 1 and 3 months last year
* The course of asthma was more than 10 years and less than 30 years
* Conform to the predetermined 4 TCM Syndrome Types
* Patients who have given written informed consent

Exclusion Criteria:

* Smoking and continuous exposure to hazardous environment
* With fever, or severity of intermittent state, high degree of sustained, or with respiratory failure, etc.
* Long term inhaled corticosteroids (more than 5 years) prior to study entry
* Pulmonary emphysema, chronic obstructive pulmonary disease, pulmonary emphysema, pulmonary heart disease, pneumonia, lung cancer and other lung diseases
* Rheumatic immune disease, diabetes, hyperthyroidism, menopause, gastroesophageal reflux, arrhythmia and other complications of the disease
* Heart, liver, kidney and other organ dysfunction
* Accompanied by other diseases of long-term use of glucocorticoids, anti allergy drugs, mental or neurological drugs or traditional Chinese Medicine
* Patients who are allergic to therapeutic medicine
* Female patients in lactation period, pregnancy or planning to get pregnant during the trial
* Patients with mental or neurological disorders

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 288 (Estimated)
Dates: Start 2017-07-30 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Asthma control rate | up to 12 months
  Asthma control rate will be measured during study of asthma at exacerbation stage within 44 days and symptom-free months will be measured on remission period within 12 months

SECONDARY OUTCOMES:
Lung function(FEV1, PVC, PEF) | up to 12 months
  Measured during study of asthma at exacerbation stage within 44 days and on remission period within 12 months
Measurement of the fractional concentration of exhaled nitric oxide | up to 12 months
  Measured during study of asthma at exacerbation stage within 44 days and on remission period within 12 months
Blood routine examination | up to 12 months
  Measured during study of asthma at exacerbation stage within 44 days and on remission period within 12 months
Cytokine levels of serum and induced sputum | up to 12 months
  Measured during study of asthma at exacerbation stage within 44 days and on remission period within 12 months
Liver function test | up to 12 months
  Measured Liver function
Kidney function test | up to 12 months
  Measured Kidney function
T cell classification | up to 12 months
  Measured T cell classification of PBMC
Cytokine levels of induced sputum | up to 12 months
  Measured cytokine levels of induced sputum supernatant

CONTACTS AND LOCATIONS:
Overall Officials: Zhenhui Lu, Doctor, Study Chair — Longhua Hospital
Locations (5):
- China (5):
  - Fenglin Street Community Health Service Center, Shanghai, Shanghai Municipality
  - Kangjian Street Community Health Service Center, Shanghai, Shanghai Municipality
  - Tianping Street Community Health Service Center, Shanghai, Shanghai Municipality
  - Longhua Hospital Affiliated Shanghai University of TCM, Shanghai, Shanghai Municipality
  - Fengxian District Hospital of TCM, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: Undecided
Through this study, to find the appropriate treatment of traditional Chinese medicine, then to further promote